CLINICAL TRIAL: NCT03573531
Title: Investigating Lipid Peroxidation Products in Donor Human Milk- a Two-Centre Pilot Study
Brief Title: Investigating Lipid Peroxidation Products in Donor Human Milk
Acronym: LIMIT
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Responsible Party: Sponsor
Other Study IDs: 1718/IRASIN/1; 221198 (Other: IRAS ID)
Record Dates: First submitted 2018-06-19; First posted 2018-06-29 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Breast Milk Collection
Keywords: donor human milk; lipid peroxidation; neonate; omega-3 fatty acids; omega-6 fatty acids; preterm infants; malondialdehyde
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Donor human milk (breast milk processed by a human milk bank)
  * Mature term breast milk
  * Preterm transitional/mature breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Donor Human Milk: Donor Human Milk (processed by a human milk bank) Sampled at two different neonatal units in the United Kingdom Collection of 5 ml of otherwise routinely discarded donor human milk
  Interventions: Other: Laboratory analysis
- Preterm Milk: Preterm transitional or mature breast milk Sampled from healthy mothers of preterm babies (born , 37 weeks gestational age) at a neonatal unit in the United Kingdom Collection of 5 ml at a time point of routine expression
  Interventions: Other: Laboratory analysis
- Term Milk: Term mature breast milk Sampled from healthy mothers of term babies in the community (e.g. Baby Cafes). Collection of 5 ml expressed for this study
  Interventions: Other: Laboratory analysis

INTERVENTIONS:
Other: Laboratory analysis — Analysis of lipid peroxidation markers (malondialdehyde, 4 hydroxy-2-nonenal, hexanal, and 8-iso-PGF2α) Analysis of fatty acid content Analysis of total antioxidant capacity

SUMMARY:
This study will quantify lipid peroxidation products (malondialdehyde, 4 hydroxy-2-nonenal, hexanal, and 8-iso-PGF2α), fatty acid content, and antioxidant capacity in donor human milk sampled from two neonatal units in the UK. Comparison will be made to preterm transitional/mature milk and term mature milk.

DETAILED DESCRIPTION:
The investigators have recently identified that current human milk banking practices in the United Kingdom may have the potential to increase levels of lipid peroxidation products in donor human milk. It is therefore important to quantify the extent of this increase. This project aims to quantify for the first time the levels of lipid peroxidation products in donor human milk that is provided to infants on the neonatal unit.

Donor human milk samples will be collected from two neonatal units in the United Kingdom, served by different human milk banks. Fresh mature term breast milk, collected from healthy mothers in the community, and preterm transitional/mature breast milk, collected from healthy mothers at a neonatal unit, will be used for comparison. For each group, 10 x 5 mL samples will be analysed for the lipid peroxidation products, malondialdehyde, 4 hydroxy-2-nonenal, hexanal, and 8-iso-PGF2α. The fatty acid content and total antioxidant capacity will also be measured. All analysis will be undertaken at Bournemouth University.

ELIGIBILITY:
Inclusion Criteria:

* Donor human milk that was intended to feed an infant at a neonatal unit in the U.K will be used for this study. Donor human milk needs to be routinely discarded 24 hours after defrosting on the unit, at that point it will be used as sample for this study.
* Preterm transitional/mature breast milk will be sampled from healthy, asymptomatic mothers of a preterm baby (born < 37 weeks gestational age) as soon as a stable milk supply is established. Samples will only be obtained if there is a surplus to the babies' need.
* Term mature breast milk will be sampled from healthy, asymptomatic mothers in the community. Samples will only be obtained if there is a surplus to the babies' need.

Exclusion Criteria:

* Donor human milk that cannot be stored on ice or in the fridge within 2 hours and cannot be frozen at -80°C within 5 hours
* For preterm and term breast milk:

Women < 18 years Women who are not able to access the study information in English Smoking women Women with mastitis Women who delivered after clinical chorioamnionitis, or other sepsis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Donor human milk is donated by mothers, having a stable milk supply, to the respective milk bank from which it is requested from the neonatal units, where it is sampled.
  Preterm mothers will be selected from a neonatal unit in the U.K.
  Term mothers will be selected from the community form baby cafes and similar in the Bournemouth area.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Lipid peroxidation markers | 2 weeks
  Analysis of malondialdehyde (TBARS, colourimetric), 4-hydroxy-2-nonenal (ELISA), hexanal (gas chromatography), and 8-iso-PGF2α (ELISA)

SECONDARY OUTCOMES:
Fatty acid content | 1 week
  Analysis of fatty acid content (gas chromatography)
Antioxidant capacity | 1 week
  Analysis of antioxidant capacity (colourimetric)

CONTACTS AND LOCATIONS:
Overall Officials: Isabell Nessel, Principal Investigator — Bournemouth University
Locations (3):
- United Kingdom (3):
  - Bournemouth University, Bournemouth
  - St George's Hospitals NHS Foundation Trust, London
  - Poole Hospital NHS Foundation Trust, Poole

REFERENCES:
- [Derived] Nessel I, De Rooy L, Khashu M, Murphy JL, Dyall SC. Long-Chain Polyunsaturated Fatty Acids and Lipid Peroxidation Products in Donor Human Milk in the United Kingdom: Results From the LIMIT 2-Centre Cross-Sectional Study. JPEN J Parenter Enteral Nutr. 2020 Nov;44(8):1501-1509. doi: 10.1002/jpen.1773. Epub 2020 Feb 11. PMID 32048312